CLINICAL TRIAL: NCT04742608
Title: Isolation and Characterization of Extracellular Vesicles in Patients With Thyroid Nodules and Thyroid Cancer
Brief Title: Development of Liquid Biopsy Technologies for Noninvasive Cancer Diagnostics in Patients With Suspicious Thyroid Nodules or Thyroid Cancer
Status: Recruiting | Type: Observational
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 19-002301; NCI-2021-00108 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 19-002301 (Other: UCLA / Jonsson Comprehensive Cancer Center)
Record Dates: First submitted 2021-02-03; First posted 2021-02-08 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-02

CONDITIONS: Thyroid Gland Carcinoma; Thyroid Gland Nodule
MeSH Terms: conditions — Thyroid Neoplasms; Thyroid Nodule

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Ancillary-correlative (biospecimen collection): Patients undergo collection of blood samples on the day of surgery following anesthesia but prior to incision and at the first routine blood test following surgery. Patients who undergo remnant ablation after total thyroidectomy with radioactive iodine have an additional blood sample collected. Patients also undergo collection of tissue samples following surgical resection of thyroid nodule or thyroid cancer. Patients' medical records are also reviewed.
  Interventions: Procedure: Biospecimen Collection; Other: Electronic Health Record Review

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood and tissue samples
Other: Electronic Health Record Review — Medical charts are reviewed

SUMMARY:
This study is being done to help researchers learn more about and successfully diagnose cancer using blood samples and tissue samples from surgeries in patients with suspicious thyroid nodules or thyroid cancer. Diagnosing cancer in this way, as opposed to biopsies, may be less invasive to the patient. Analyzing blood and tissues samples may also help researchers to differentiate non-cancerous tumors from thyroid cancer and detect high-risk mutations to guide treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Sensitivity and specificity of molecular profile of thyroid derived extracellular vesicles (EVs) as predictor of thyroid cancer.

SECONDARY OBJECTIVES:

I. Quantity of thyroid derived EVs captured in various stages of thyroid cancer.

II. Whether quantity of EVs decreases in proportion to response to therapy in thyroid cancer patients.

III. Optimal ribonucleic acid (RNA)/deoxyribonucleic acid (DNA) panel in thyroid tumor derived EVs to diagnose thyroid cancer.

OUTLINE:

Patients undergo collection of blood samples on the day of surgery following anesthesia but prior to incision and approximately 4-6 weeks after surgery. Patients who undergo remnant ablation after total thyroidectomy with radioactive iodine have an additional blood sample collected. Patients also undergo collection of tissue samples following surgical resection of the thyroid. Patients' medical records are also reviewed.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 and older
* Consented for thyroid surgery for thyroid cancer or indeterminate thyroid nodule

Exclusion Criteria:

* Patients with concurrent malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in endocrine surgery clinic sites across University of California, Los Angeles (UCLA) who have undergone thyroid fine needle aspiration biopsy.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2020-02-21 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of molecular profile of thyroid-derived extracellular vesicles | Up to 3 years
Specificity of molecular profile of thyroid-derived extracellular vesicles | Up to 3 years
Negative predictive value of molecular profile of thyroid-derived extracellular vesicles | Up to 3 years
Positive predictive value of molecular profile of thyroid-derived extracellular vesicles | Up to 3 years

SECONDARY OUTCOMES:
Quantity of thyroid-derived extracellular vesicles captured in patients with localized, regional, and distant disease versus benign thyroid adenomas | Up to 3 years
Quantity of thyroid-derived extracellular vesicles captured in patients with excellent, indeterminate, biochemically incomplete, and structural incomplete responses to initial therapy | Up to 3 years
Combination of ribonucleic acid/deoxyribonucleic acid-based tests that can be perf thyroid-derived extracellular vesicles | Up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: James Wu, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (1):
- UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No